CLINICAL TRIAL: NCT03356977
Title: A PHASE 4, MULTICENTER, OPEN-LABEL SAFETY STUDY OF CRISABOROLE OINTMENT 2% IN CHILDREN AGED 3 MONTHS TO LESS THAN 24 MONTHS WITH MILD TO MODERATE ATOPIC DERMATITIS
Brief Title: A Study of Crisaborole Ointment 2% in Children Aged 3-24 Months With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3291002; CARE 1 (Other: Alias Study Number)
Record Dates: First submitted 2017-10-31; First posted 2017-11-29 (Actual); Results first posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — crisaborole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Crisaborole ointment 2% (Experimental): Subjects will be dosed for 28 days. A thin layer of ointment will be applied to all areas designated for treatment.
  Interventions: Drug: Crisaborole ointment 2%

INTERVENTIONS:
Drug: Crisaborole ointment 2% — Applied BID
  Other Names: Eucrisa

SUMMARY:
This 4-week study will evaluate the safety, pharmacokinetics (PK), and efficacy of crisaborole ointment 2%, applied twice daily (BID) in subjects who are 3 months to less than 24 months of age with mild-to-moderate AD.

DETAILED DESCRIPTION:
Approximately 125 subjects will be enrolled. Subjects must have mild-to-moderate AD involving at least 5% treatable %BSA assessed on Baseline/Day 1. Treatable %BSA will be defined as the percent of a subject's total body surface area that is AD-involved, excluding the scalp.

In addition, a cohort of at least 16 of the 125 subjects will be included in a subgroup for PK assessment. These subjects must have moderate AD and a minimum of 35% treatable %BSA, excluding the scalp, and must complete all PK assessments to be included in the PK analysis. Of these subjects, at least 3 subjects who are less than 9 months of age will be enrolled. Subjects discontinuing for reasons other than treatment emergent adverse event ( TEAE) may be replaced at the discretion of the sponsor to ensure 16 subjects complete the PK assessments. Only selected study sites will participate in the PK assessment.

Scheduled study visits/telephone contacts for all subjects will occur at Screening (up to 28 days prior to Baseline/Day 1), Baseline/Day 1, Day 8, Day 15, Day 22, Day 29 (end of treatment/early termination), Day 36, and Day 57 (end of study).

ELIGIBILITY:
Inclusion Criteria:

Aged ≥ 3 months at the screening visit to < 24 months on baseline/Day 1, diagnosed with AD

Exclusion Criteria:

Subjects with any clinically significant dermatological condition or disease (including active or potentially recurrent non-AD dermatological conditions that overlap with AD such as Netherton Syndrome)

Ages: 3 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- United States (23):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Rady Children's Hospital - San Diego/University of California, San Diego, San Diego, California
  - Rady Children's Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - IMMUNOe Research Centers, Thornton, Colorado
  - Baumann Cosmetic and Research Institute, Miami, Florida
  - DS Research, Louisville, Kentucky
  - Craig A. Spiegel, M.D., Bridgeton, Missouri
  - Skin Specialists, PC, Omaha, Nebraska
  - Ohio Pediatric Research Association, Inc., Dayton, Ohio
  - Oklahoma State University - Center for Health Sciences, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - DermResearch, Inc., Austin, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Tanner Clinic, Layton, Utah
  - Jordan Valley Dermatology Center, West Jordan, Utah
  - Timber Lane Allergy & Asthma Research, LLC, South Burlington, Vermont
  - PI-Coor Clinical Research, LLC, Burke, Virginia
  - Pediatric Associates of Charlottesville, PLC, Charlottesville, Virginia
  - Pediatric Research of Charlottesville, LLC (Regulatory Only), Charlottesville, Virginia
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
  - Dermatology Specialists of Spokane, Spokane, Washington
- Australia (6):
  - Australian Clinical Research Network Pty Ltd, Maroubra, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Eastern Health, Box Hill, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - The Royal Children's Hospital, Parkville, Victoria
- Canada (3):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Lynderm Research Inc., Markham, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Schlessinger J, Shepard JS, Gower R, Su JC, Lynde C, Cha A, Ports WC, Purohit V, Takiya L, Werth JL, Zang C, Vlahos B; CARE 1 Investigators. Safety, Effectiveness, and Pharmacokinetics of Crisaborole in Infants Aged 3 to < 24 Months with Mild-to-Moderate Atopic Dermatitis: A Phase IV Open-Label Study (CrisADe CARE 1). Am J Clin Dermatol. 2020 Apr;21(2):275-284. doi: 10.1007/s40257-020-00510-6. PMID 32212104
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3291002

RESULTS

PARTICIPANT FLOW:
Groups:
- Crisaborole Topical Ointment, 2 Percent: Participants with mild to moderate atopic dermatitis (AD) received crisaborole ointment, 2 percent on treatable AD lesions, twice daily from Day 1 to Day 29. Treatable AD lesions were identified at Baseline (Day 1) by investigator.
Period: Overall Study
Arm/Group | Crisaborole Topical Ointment, 2 Percent
Started | 137
Completed | 132
Not Completed | 5
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by parent/guardian | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set included any participant who received at least 1 dose of investigational product.
Groups:
- Crisaborole Topical Ointment, 2 Percent: Participants with mild to moderate AD received crisaborole ointment, 2 percent on treatable AD lesions, twice daily from Day 1 to Day 29. Treatable AD lesions were identified at Baseline (Day 1) by investigator.
Arm/Group | Crisaborole Topical Ointment, 2 Percent
Number analyzed (Participants) | 137
Age, Continuous [Mean (Standard Deviation); unit: months] | 13.6 (6.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 118
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 27
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 11
  White | 84
  More than one race | 13
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs), Serious Adverse Events (SAEs) and Site Reactions
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. Treatment-emergent were events between first dose of investigational product and up to 28 days after the last dose of investigational product that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs. Site reactions are reactions which occurred in participants at the site of application of investigational product.
Time Frame: Baseline (Day 1) up to at least 28 days after last dose of investigational product (up to 60 days)
Population: Safety analysis set included any participant who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Crisaborole Topical Ointment, 2 Percent
Number analyzed (Participants) | 137
Participants
  AEs | 88
  SAEs | 1
  Application site Reactions | 15

2. Primary Outcome: Number of Participants With Clinically Significant Height Values Meeting Pre-defined Criteria
Description: Height of participants was measured in terms of centimeter (cm). The pre-defined criteria for measuring the height was less than (<) 55 cm and greater than (>) 92.5 cm.
Time Frame: Baseline (Day 1) up to Day 29 (end of treatment)
Population: Safety analysis set included any participant who received at least 1 dose of investigational product. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Crisaborole Topical Ointment, 2 Percent
Number analyzed (Participants) | 134
Participants
  < 55 cm | 0
  > 92.5 cm | 3

3. Primary Outcome: Number of Participants With Clinically Significant Weight Values Meeting Pre-defined Criteria
Description: Weight of participants was measured in terms of kilogram (kg). The pre-defined criteria of measuring the weight of participants was less than equal to (<=) 4.5 kg and >15 kg.
Time Frame: Baseline (Day 1) up to Day 29 (end of treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Crisaborole Topical Ointment, 2 Percent
Number analyzed (Participants) | 135
Participants
  <= 4.5 kg | 0
  > 15 kg | 3

4. Primary Outcome: Number of Participants With Clinically Significant Blood Pressure Values Meeting Pre-defined Criteria
Description: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) of participants was measured in terms of millimeters of mercury (mmHg). The clinically significant pre-defined criteria were, SBP: change of greater than equal to (>=) 30 mmHg increase from baseline (IFB) and SBP change of >= 30 mmHg decrease from baseline (DFB); DBP: change of >=20 mmHg IFB and DBP change of >=20 mmHg DFB.
Time Frame: Baseline (Day 1) up to Day 29 (end of treatment)
Population: Safety analysis set included any participant who received at least 1 dose of investigational product. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants evaluable for specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Crisaborole Topical Ointment, 2 Percent
Number analyzed (Participants) | 136
Participants
  SBP:change of>=30 mmHg IFB | 3
  SBP:change of>=30 mmHg DFB | 4
  DSBP: change of >= 20 mmHg IFB: number analyzed (Participants) | 135
  DSBP: change of >= 20 mmHg IFB | 8
  DSBP: change of >= 20 mmHg DFB: number analyzed (Participants) | 135
  DSBP: change of >= 20 mmHg DFB | 18

5. Primary Outcome: Number of Participants With Clinically Significant Pulse Rate Values Meeting Pre-defined Criteria
Description: Pulse rate of participants was measured in terms of beats per minute (bpm). The pre-defined criteria of measuring the pulse rate of participants was <90 bpm and >180 bpm.
Time Frame: Baseline (Day 1) up to Day 29 (end of treatment)
Population: Safety analysis set included any participant who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Crisaborole Topical Ointment, 2 Percent
Number analyzed (Participants) | 137
Participants
  <90 bpm | 12
  >180 bpm | 0

6. Primary Outcome: Number of Participants With Clinically Significant Respiratory Rate Values Meeting Pre-defined Criteria
Description: Respiratory rate was measured in terms of number of breaths per minute. The pre-defined criteria of measuring the respiratory rate of participants was < 22 breaths per min and > 53 breaths per min.
Time Frame: Baseline (Day 1) up to Day 29 (end of treatment)
Population: Safety analysis set included any participant who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Crisaborole Topical Ointment, 2 Percent
Number analyzed (Participants) | 137
Participants
  < 22 breaths per minute | 17
  > 53 breaths per minute | 4

7. Primary Outcome: Number of Participants With Clinically Significant Body Temperature Values Meeting Pre-defined Criteria
Description: Body temperature of participants was measured in degree Celsius. The normal body temperature value was >= 39 degree Celsius.
Time Frame: Baseline (Day 1) up to Day 29 (end of treatment)
Population: Safety analysis set included any participant who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Crisaborole Topical Ointment, 2 Percent
Number analyzed (Participants) | 137
Participants | 0

8. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Values Meeting Pre-defined Criteria
Description: ECG of participants was measured in terms of millisecond (msec). ECG parameters included pulse rate (PR) interval, QRS interval, corrected QT interval using Fridericia's formula (QTcF). ECG values meeting pre-defined criteria were 1) PR interval: greater than equal to (>=) 25 percent (%) increase when baseline greater than (>)200 milliseconds (msec); or increase >=50% when baseline less than or equal to (<=200) msec; 2) QRS interval: >=25% increase when baseline >100 msec; >=50% increase when baseline <= 100 msec; 3) QTCF interval: QTc interval using Fridericia's formula (QTcF interval) > 30 msec. IFB stands for increase from baseline.
Time Frame: Baseline (Day 1) up to Day 29 (end of treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Crisaborole Topical Ointment, 2 Percent
Number analyzed (Participants) | 135
Participants
  PR Interval: > 200 msec and >=25% IFB | 0
  PR Interval: <= 200 msec and >=50% IFB | 1
  QRS Duration: >= 100 msec and >= 25% IFB | 0
  QRS Duration: < 100 msec and >= 50% IFB | 0
  QTcF Interval: >30 msec | 10

9. Primary Outcome: Number of Participants With Clinically Significant Laboratory Parameters Meeting Pre-defined Criteria
Description: Criteria: hematology: hemoglobin, hematocrit, erythrocytes < 0.8*lower limit of normal (LLN), platelets <0.5*LLN >1.75*upper limit of normal (ULN), leukocytes <0.6* LLN >1.5* ULN, lymphocytes, lymphocytes/leukocytes, neutrophils, neutrophils/leukocytes <0.8* LLN >1.2* ULN, basophils, basophils/leukocytes, eosinophils, eosinophils/leukocytes monocytes monocytes/leukocytes >1.2*ULN. Clinical chemistry: bilirubin >1.5*ULN, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase >3.0*ULN, protein, albumin <0.8* LLN >1.2* ULN, blood urea nitrogen, creatinine >1.3* ULN, sodium <0.95*LLN >1.05*ULN, potassium, chloride, bicarbonate <0.9* LLN >1.1* ULN, glucose <0.6*LLN >1.5*ULN.
Time Frame: Baseline (Day 1) up to Day 29 (end of treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Crisaborole Topical Ointment, 2 Percent
Number analyzed (Participants) | 122
Participants | 105

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to at least 28 days after last dose of investigational product (up to 60 days)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Crisaborole Topical Ointment, 2 Percent
All-Cause Mortality (participants affected / at risk) | 0/137
Serious Adverse Events (participants affected / at risk) | 1/137
Other Adverse Events (participants affected / at risk) | 41/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crisaborole Topical Ointment, 2 Percent (N=137)
Febrile convulsion (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crisaborole Topical Ointment, 2 Percent (N=137)
Diarrhoea (Gastrointestinal disorders) | 10
Pyrexia (General disorders) | 13
Upper respiratory tract infection (Infections and infestations) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 9
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT03356977/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT03356977/SAP_001.pdf